CLINICAL TRIAL: NCT06359288
Title: Effect of QR Code Supported Infant Care Training Given to Preterm Newborn Mothers on Motherhood Self-Efficacy and Anxiety
Brief Title: Preterm Newborn Mothers' Anxiety and Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Sinem Yalnızoglu Caka, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023/01.11/2023/6
Record Dates: First submitted 2024-04-02; First posted 2024-04-11 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Nursing Care; Mother-Infant Interaction; Education
Keywords: Motherhood Self-Efficacy; Anxiety; Nursing Care; Preterm; QR code
MeSH Terms: conditions — Anxiety Disorders; Premature Birth

STUDY DESIGN:
Intervention Model Description: The study was conducted experimentally with a pre-test and post-test control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinding was used in the study. For this purpose, the participants were not specified in which group they belonged to the research. Therefore, a separate informed consent form was prepared for each group. In order to avoid bias in the analysis of the research data, statistician blinding was also applied.
  While coding the research data, the research groups were coded as A and B, and the statistician was prevented from knowing which letter represented which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving QR code supported training (Experimental): Training sessions in the training class run three days a week for two weeks. 6. During the training process, QR codes were integrated into the sections related to the care of the newborn in the guide in order to provide mothers with the opportunity to watch the video simultaneously while reading the guide in practices requiring skills related to hygienic care of the newborn and nutrition / communication / sleep, and to allow them to watch it repeatedly as long as they feel the need. In these videos, the application steps were shown one by one. URL addresses of the videos were obtained and then QR Codes were created. When the code is scanned with a smartphone, it automatically redirects the user to the specified URL. The difference between the groups was that videos on newborn care were shown and QR Code training guides with the same content as the SC group created by the researchers on newborn care were distributed.
  Interventions: Other: Group receiving QR code supported training
- Recommendations to start care (No Intervention): In the training class, mothers who are preparing for discharge are currently given training on the appearance, feeding, care, vaccinations, sleep and health checks of the premature infant, and the care of the newborn is carried out practically.

INTERVENTIONS:
Other: Group receiving QR code supported training — During the training process, QR codes were integrated into the sections related to the care of the newborn in the guide to provide mothers with the opportunity to watch the video simultaneously while reading the guide in practices requiring skills related to hygienic care of the newborn and nutrition / communication / sleep, and to allow them to watch it repeatedly as long as they feel the need. In these videos, the application steps were shown one by one. When the code is scanned with a smartphone, it automatically redirects the user to the specified URL. The QR codes in the Implementation Guide on the Care of the Newborn consist of eight videos) that allow mothers to watch the hygienic care of the newborn in practice. After the end of this phase of the training, the questionnaires were re-administered to the mothers in both groups one month after discharge.
  Arms: Group receiving QR code supported training

SUMMARY:
The aim of this study was to evaluate the effect of QR code supported infant care training given to mothers of preterm newborns on maternal self-efficacy and maternal anxiety level .

DETAILED DESCRIPTION:
Maternal and child health is an important health indicator of societies. According to the World Health Organisation, almost half of all under-five child deaths are neonatal deaths. In order to reduce these deaths, especially in the neonatal period, it is very important for mothers to learn and correctly apply infant care. In studies conducted with mothers of preterm newborns, it was determined that mothers felt themselves inadequate after taking care responsibilities after discharge, expressed that they needed training for the care of the baby, and preferred to remain bystanders because they were less confident in the care of the baby. However, other studies have reported that preterm and hospitalised infants have a negative impact on the development of the mothering role. Prematurity may increase maternal anxiety and negatively affect perceived maternal self-efficacy. At the same time, the mother's intense anxiety and inadequate perceived maternal self-efficacy negatively affect infant care.

Maternal self-efficacy perception is mothers' beliefs about being successful in their parenting role and is an important mechanism guiding the interactions of preterm newborns and their mothers in the hospital. In order for this mechanism to continue in a healthy way, the nurse should identify the aspects that mothers perceive themselves as adequate or that mothers perceive as negative from birth and observe all their interventions towards the baby. Self-efficacy, which can be gained through learning by observation, can be maximised in the postnatal period by nurses demonstrating the principles they want to teach. Therefore, nurses should clearly show the practices for infant care to mothers and support the perception of maternal self-efficacy.

Today, traditional materials used in the educational process (blackboard, book, etc.) are replaced by smart and portable devices (e-book, smart board, tablet, etc.). In this context, QR codes serve as a bridge between old and new education models. In other words, QR codes increase the effectiveness of mobile education by integrating mobile devices into traditional educational materials. QR codes are a cheap and easy process for delivering information to individuals. When the literature is analysed, it is seen that the interest and motivation in the subject increases when the training sessions offered through the internet and printed learning materials are used together. QR codes are frequently used in educational activities due to their versatility and their ability to enable different learning environments. When the benefits of QR codes are analysed in studies conducted on healthcare professionals, students, and educators in the literature, they can be listed as ease of use and ease of access, adaptability, simplicity of development and potential environmental benefits compared to other access methods. However, studies on the use of QR codes in patient education in the field of nursing are limited.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infant who were born between 28-36+6 gestational weeks
* Preterm infant with a low birth weight at hospitalization (between 1500-2500 g)
* Preterm infant weight of 2500 g or more at discharge,
* Preterm infant who had stable vital signs,
* Preterm infant who do not use muscle relaxants, analgesics, sedatives or inotropic drugs,
* Preterm infant who do not have a serious neurological disease
* Mothers who stay with the baby for at least one month after discharge,
* Mothers who voluntarily accepting the study,
* Mothers who not being diagnosed with a psychiatric illness.

Exclusion Criteria:

* Mothers who did not have the ability to read and understand Turkish,
* Mothers who did not use/access the internet,
* Mothers who had twin babies
* Mothers whose babies with a disease that would prevent post-discharge care

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Must be biological mother
Enrollment: 80 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-03-23 (Actual)

PRIMARY OUTCOMES:
Perceived Maternal Self-Efficacy Scale (PMES)- Survey | Before the recruit pre-test (PMES- survey scale) will be applied. One months after the intervention post-test (PMES survey scale) again will be applied.
  QR code-supported education given to mothers of preterm newborns improves. The scale assesses the perceived maternal self-efficacy levels of mothers of hospitalised preterm infants. The scale, which consisted of 19 items, was graded between 1 and 4 (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree). Scoring of the scale was calculated by adding the obtained scores. The score obtained from the scale is between 19 and 76. A high score indicates that the mother's self-efficacy is high. The reliability coefficient of the scale in mothers of hospitalised preterm infants was 0.98. In this study, the internal consistency coefficient of the scale was found to be 0.95.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI)- Survey Scale | Before the recruit pre-test (STAI- survey scale) will be applied. One months after the intervention post-test (STAI survey scale) again will be applied.
  QR code-supported education given to mothers of preterm newborns decreases the mother's anxiety level.The STAI provides information about state anxiety. The STAI consists of 20 items and is graded between 1-4 according to the anxiety level of the person. The scale includes plain and inverted statements (items: 1., 2., 5., 8., 10., 11., 15., 16., 19. and 20.) determining positive and negative emotions. Scores between 20-80 are obtained from the scale. A higher score means higher anxiety. In scoring, the total score of the negative statements is subtracted from the total score of the positive statements. A predetermined and unchanged 50 points are added to this score. The score obtained indicates the anxiety level of the person. In this study, the internal consistency coefficient of the scale was found to be 0.88.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, İzmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellot J, Shaffer K, Wang M. Use of quick response coding to create interactive patient and provider resources. J Nurs Educ. 2015 Apr;54(4):224-7. doi: 10.3928/01484834-20150318-07. PMID 25826764
- [Background] Barnes CR, Adamson-Macedo EN. Perceived Maternal Parenting Self-Efficacy (PMP S-E) tool: development and validation with mothers of hospitalized preterm neonates. J Adv Nurs. 2007 Dec;60(5):550-60. doi: 10.1111/j.1365-2648.2007.04445.x. PMID 17973719
- [Background] Afand N, Keshavarz M, Fatemi NS, Montazeri A. Effects of infant massage on state anxiety in mothers of preterm infants prior to hospital discharge. J Clin Nurs. 2017 Jul;26(13-14):1887-1892. doi: 10.1111/jocn.13498. Epub 2017 Mar 24. PMID 27486850
- [Background] Kadiroglu T, Guducu Tufekci F. Effect of Infant Care Training on Maternal Bonding, Motherhood Self-Efficacy, and Self-Confidence in Mothers of Preterm Newborns. Matern Child Health J. 2022 Jan;26(1):131-138. doi: 10.1007/s10995-021-03287-0. Epub 2021 Nov 27. PMID 34837599
- [Background] Pazarcıkcı F, Efe E. (2017). Preterm Bebeklerin Taburculuk Sonrası Evde Bakımının Sağlanmasında Hemşirenin Rolü. MAKÜ Sag. Bil. Enst. Derg, 5 (1), 45-52.
- [Background] Pisoni C, Garofoli F, Baiardini I, Tzialla C, Stronati M. The development of parents-infant relationship in high-risk pregnancies and preterm birth. JPNIM, 2014, 3: e030233.
- [Background] Rawlins LN, Seaman KA. The Use of QR Codes to Engage Nursing Students With Next Generation NCLEX. J Nurs Educ. 2024 Mar;63(3):186-187. doi: 10.3928/01484834-20240108-02. Epub 2024 Mar 1. PMID 38442404
- [Background] Ritchie SK. Primary care of the premature infant discharged from the neonatal intensive care unit. MCN Am J Matern Child Nurs. 2002 Mar-Apr;27(2):76-85. doi: 10.1097/00005721-200203000-00004. PMID 11984275
- [Background] Shorey S, Chan SW, Chong YS, He HG. Maternal parental self-efficacy in newborn care and social support needs in Singapore: a correlational study. J Clin Nurs. 2014 Aug;23(15-16):2272-82. doi: 10.1111/jocn.12507. Epub 2013 Dec 26. PMID 24372630
- [Background] Tognasso G, Gorla L, Ambrosini C, Figurella F, De Carli P, Parolin L, Sarracino D, Santona A. Parenting Stress, Maternal Self-Efficacy and Confidence in Caretaking in a Sample of Mothers with Newborns (0-1 Month). Int J Environ Res Public Health. 2022 Aug 5;19(15):9651. doi: 10.3390/ijerph19159651. PMID 35955005
- [Background] Wolke D, Eryigit-Madzwamuse S, Gutbrod T. Very preterm/very low birthweight infants' attachment: infant and maternal characteristics. Arch Dis Child Fetal Neonatal Ed. 2014 Jan;99(1):F70-5. doi: 10.1136/archdischild-2013-303788. Epub 2013 Jun 21. PMID 23792355
- [Background] Yayan, E. H., Özdemir, M., Düken, M. E., Suna Dağ, Y. (2019). Yenidoğan Yoğun Bakım Ünitesinde Bebeği Yatan Ebeveynlerin Stres Düzeylerinin Belirlenmesi, Gümüşhane Üniversitesi Sağlık Bilimleri Dergisi (GÜSBD), 8(1), 82-89.
- [Background] Shrestha S, Adachi K, Petrini MA, Shrestha S, Rana Khagi B. Development and evaluation of a newborn care education programme in primiparous mothers in Nepal. Midwifery. 2016 Nov;42:21-28. doi: 10.1016/j.midw.2016.09.006. Epub 2016 Sep 15. PMID 27710817
- [Background] Silva, I. O. A. M. D., Aredes, N. D. A., Bicalho, M. B., Delácio, N. C. B., Mazzo, L. D. L., & Fonseca, L. M. M. (2018). Booklet on premature infants as educational technology for the family: quasi-experimental study. Acta Paulista de Enfermagem, 31, 334-341. https://doi.org/10.1590/1982-0194201800048
- [Derived] Caka SY, Topal S, Ozturkler S, Celenkoglu FT, Gunlemez A. The Effect of QR Code Supported Newborn Care Training Given to Mothers With Premature Infant on Self-Efficacy and Anxiety: A Randomised Controlled Study. Scand J Caring Sci. 2025 Sep;39(3):e70051. doi: 10.1111/scs.70051. PMID 40605472